CLINICAL TRIAL: NCT07158437
Title: A Randomized, Double-Blind, Placebo-Controlled Single-Ascending Dose and Multiple-Ascending Dose Phase 1 Study of SL-325 in Healthy Volunteers
Brief Title: Phase 1 Study of SL-325 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shattuck Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SL-325-101
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: DR3; SL-325
MeSH Terms: interventions — 3-(2-(4-quinolin-3-yl)benzyl-1-oxoisoindolin-6-yl)-N-hydroxy-acrylamide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAD: SL-325 (Experimental): Participants will receive a single dose of SL-325 in escalating dose cohorts
  Interventions: Biological: SL-325
- SAD: Placebo (Placebo Comparator): Participants will receive a single dose of placebo (normal saline)
  Interventions: Other: Placebo (Normal Saline)
- MAD: SL-325 (Experimental): Participants will receive a three doses of SL-325 in escalating dose cohorts
  Interventions: Biological: SL-325
- MAD: Placebo (Placebo Comparator): Participants will receive a three doses of placebo (normal saline)
  Interventions: Other: Placebo (Normal Saline)

INTERVENTIONS:
Biological: SL-325 — DR3 blocking antibody
  Arms: MAD: SL-325; SAD: SL-325
Other: Placebo (Normal Saline) — Normal saline
  Arms: MAD: Placebo; SAD: Placebo

SUMMARY:
This first-in-human study is a randomized, double-blind, placebo-controlled, single-ascending dose and multiple-ascending dose study of SL-325 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent
2. 18-55 years of age, inclusive, at the time of signing the informed consent form
3. Body mass index of 18-32 kg/m2, inclusive, and a total body weight > 50 kg
4. Laboratory values within normal limits or any abnormalities deemed not clinically significant by the Investigator
5. Participant agrees to practice birth control measures

Exclusion Criteria:

1. History or presence of a clinically significant infectious disease or hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, neurologic, or psychiatric abnormality
2. Any clinically significant abnormality on vital signs, electrocardiogram (ECG), or laboratory parameters
3. History of regular alcohol consumption within 6 months of Screening
4. Positive test for use of drugs or alcohol at Screening
5. History of use of tobacco- or nicotine-containing products within 3 months of Screening
6. History of infusion-related reaction or allergic reaction upon receipt of an IV infusion
7. Positive hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV) test at Screening
8. Blood donation within 90 days prior to Day -1 or plasma donation within 1 week prior to Day 1
9. Receipt of specific medications within a specified time period
10. Women who are currently breastfeeding or have a positive pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Day 1 through 75 days after last dose
  Incidence and severity of treatment-emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Cmax | Day 1 through 75 days after last dose
  Maximum observed concentration
Pharmacokinetics (PK): Tmax | Day 1 through 75 days after last dose
  Time at which the maximum concentration is observed
Pharmacokinetics (PK): Ctrough | Day 1 through 75 days after last dose
  Minimum observed concentration following a single dose
Pharmacokinetics (PK): AUC | Day 1 through 75 days after last dose
  Area under the concentration-time curve
Pharmacokinetics (PK): T1/2 | Day 1 through 75 days after last dose
  Terminal elimination half-life
Pharmacokinetics (PK): CL | Day 1 through 75 days after last dose
  Clearance
Pharmacokinetics (PK): Vz | Day 1 through 75 days after last dose
  Volume of distribution
Immunogenicity: Number/proportion of participants with positive or negative anti-drug antibody (ADA) titers | Day 1 through 75 days after last dose
Immunogenicity: Number/proportion of participants with neutralizing anti-drug antibodies | Day 1 through 75 days after last dose
Immunogenicity: Time to onset and duration of anti-drug antibodies | Day 1 through 75 days after last dose
Immunogenicity: Number/proportion of participants with transient vs persistent anti-drug antibodies | Day 1 through 75 days after last dose
Receptor Occupancy: Percent of DR3-positive T cells bound by SL-325 | Day 1 through 75 days after last dose
Receptor Occupancy: Duration of DR3-positive T cell binding by SL-325 | Day 1 through 75 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No